CLINICAL TRIAL: NCT05458349
Title: Acellular Dermis in Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROH11ORTH09
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries
Keywords: rotator cuff; shoulder; surgery; acellular dermal graft; acellular dermis; rotator cuff augmentation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: It is a Level 1 study, a prospective double blind, randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dermis group (Experimental): Group will receive standard of care treatment and interventions plus the use of the acellular dermal graft during surgery
  Interventions: Device: acellular dermis
- control group (No Intervention): Group will receive standard of care treatment and interventions but the acellular dermal graft will not be used during surgery

INTERVENTIONS:
Device: acellular dermis
  Arms: dermis group

SUMMARY:
To determine if an acellular dermal graft (ADG) will incorporate into the rotator cuff and subsequently improve outcomes without an increase in risk to the patient

DETAILED DESCRIPTION:
Rotator cuff healing poses a significant clinical problem with re-tear rates between 20-50%. The final functional outcome following surgery correlates with healing, with those that completely heal performing best. Failure of repair is mainly due to tendon failure both mechanically and biologically. If the healing and the structural properties of the tendon can be improved then significant functional gains may be achieved. This study will therefore utilise acellular dermal grafts to determine whether they could be used for to improve patient outcomes following surgery

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic rotator cuff tear that warrants operative intervention.
2. A Tear measuring between 1-5cm at arthroscopy.
3. An arthroscopic rotator cuff repair.
4. Written consent.

Exclusion Criteria:

1. Rotator cuff tears greater than 5cm and less than 1cm
2. Clinical or radiological evidence of osteoarthritis affecting the index side.
3. Patients involved in a Compensation claim related to the shoulder.
4. Inability to attend follow-up for 1 year and to a repeat MRI scan.
5. Previous shoulder surgery or proximal humeral fracture on the index side.
6. Patients that are recruited in a current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
rotator cuff healing | 12 month post-surgery
  Rotator cuff healing on MRI

SECONDARY OUTCOMES:
Western Ontario Rotator cuff score | 12months
  comparison of scores between groups
Constant Murley score | 12 months
  comparison of scores between groups
American shoulder and elbow surgeons standardized form | 12 months
  comparison of scores between groups

CONTACTS AND LOCATIONS:
Overall Officials: Martyn Mr Snow, MD, Principal Investigator — The Royal Orthopaedic Hospital NHS Foundation Trust
Locations (1):
- The Royal Orthopaedic Hospital NHS Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No